CLINICAL TRIAL: NCT03377881
Title: STHLM3 MR Phase 2: A New Diagnostic Chain for Prostate Cancer Detection Using the Stockholm3 Test and MR/Fusion Biopsies
Brief Title: Prostate Cancer Detection Using the Stockholm3 Test and MR/Fusion Biopsies
Acronym: STHLM3MR-2
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Tobias Nordström, Urologist PhD Principal Investigator, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: STHLM3MR-2
Record Dates: First submitted 2017-11-28; First posted 2017-12-19 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Two-step design with a first step using paired design for blood-analysis and a second step using randomisation between prostate biopsy strategy. Repeated screening using individualised screen intervals for participants randomised to the experimental (MRI) arm and without prostate cancer diagnosed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard arm (One testing with PSA and standard biopsy) (Other): The traditional/control arm consists of PSA testing and if PSA>3ng/ml a systematic biopsy of the prostate is performed. Only one screening is offered for participants.
  Interventions: Procedure: Systematic biopsies
- STHLM3+MRI/Fusion including repeat screening. (Experimental): The experimental arm consists of a Stockholm3 bloodiest and if elevated, an MRI is recommended with targeted biopsies to prostate lesions. Participants with PSA<1.5ng/ml are reinvented for prescreen after 6 years. Remaining participants with no prostate cancer detected are reinvited for re-screen at 2-3 years.
  Interventions: Procedure: MRI/Fusion biopsies

INTERVENTIONS:
Procedure: MRI/Fusion biopsies — The intervention in the experimental arm is an MRI with targeted biopsies using fusion technique to prostate lesions. Repeat screening is offered after 2-6 years on an individualised basis.
  Arms: STHLM3+MRI/Fusion including repeat screening.
Procedure: Systematic biopsies — The intervention in the control arm is traditional systematic biopsies of the prostate.
  Arms: Standard arm (One testing with PSA and standard biopsy)

SUMMARY:
The STHLM3-MRI trial is a study comparing traditional prostate cancer detection using PSA and systematic biopsies with the improved pipeline for prostate cancer detection using the STHLM3 test and targeted biopsies in a screening context.

The study includes individualised repeat invitations for re-screening to participants not diagnosed with prostate cancer.

DETAILED DESCRIPTION:
The overarching strategy of the STHLM3-MR/Fusion projects are to study an improved diagnostic pipeline including an improved blood-based test for identification of men with increased risk of prostate cancer and use of MRI to select men for diagnostic workup with targeted prostate biopsies. The aim is to increase the specificity in early detection of prostate cancer without decreasing the sensitivity of aggressive prostate cancers.

The primary endpoints are the number of performed biopsies, the number of performed MRI and the number of detected high-risk prostate cancers. Secondary endpoints include the number of low risk prostate cancers diagnosed and the proportion of patients with up-or downgraded disease after assessment of prostatectomy specimen. Additional aims include to assess the health economic consequences and development of automated image-analysis.

The STHLM3-MR project is performed in two separate phases, analyzed separately. STHLM3-MR Phase 1 closed inclusion 2017-06-01. All participants underwent target and systematic biopsies together with STHLM3 test analysis. The study is constitutes a current practice cohort and levels of the STHLM3 test were not used for selecting participants.

STHLM3-MR Phase 2 is a study comparing traditional prostate cancer detection using PSA and systematic biopsies with the improved pipeline for prostate cancer detection using the STHLM3 test and targeted biopsies in a screening context. STHLM3-MR Phase 2 reported outcomes from the first screening round 2023. Repeated screening with individualised screening intervals will be offered to participants without prostate cancer detected.

ELIGIBILITY:
Inclusion Criteria:

* Permanent postal address in Stockholm

Exclusion Criteria:

* • Severe illnesses such as metastatic cancers, severe cardio-vascular disease or dementia

  * Contraindications for magnetic resonance imaging (MRI) eg pacemaker, magnetic cerebral clips, cochlear implants or severe claustrophobia.

Ages: 50 Years to 74 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12750 (Actual)
Dates: Start 2018-04-04 (Actual); Primary Completion 2020-12-10 (Actual); Study Completion 2030-12-10 (Estimated)

PRIMARY OUTCOMES:
Number of detected cancers characterized as Gleason Score ≥7 on evaluation of biopsy specimen | At 2 months after completing first screening round (included biopsy procedure). At two months after completing repeat screening rounds ( year 3, 6, 9, 12 and 15).
  Cancers detected by pathological evaluation of biopsy specimen collected from the respective study arm

SECONDARY OUTCOMES:
Number of detected cancer with Gleason Score 6 | At 2 months after completing first screening round (last included biopsy procedure). At two months after completing repeat screening rounds ( year 3, 6, 9, 12 and 15).
  Cancers detected by pathological evaluation of biopsy specimen collected from the respective study arm
Number of performed biopsy procedures in the study arms | At 2 months after completing first screening round (last included biopsy procedure). At two months after completing repeat screening rounds ( year 3, 6, 9, 12 and 15).
  Number of performed prostate biopsy procedures counted per study arm
Number of performed MRI in the study arms | At 2 months after completing first screening round (last included biopsy procedure). At two months after completing repeat screening rounds ( year 3, 6, 9, 12 and 15).
  Number of performed prostate MRI procedures counted per study arm
Number of infectious complications | Questionnaire collection finalised within 2months after last biopsy procedure in study
  As assessed by questionnaire within 2 month after biopsy procedure
Distribution of MRI findings in men positive for Stockholm3 and/or PSA | At 2 months after completing first screening round (last included biopsy procedure). At two months after completing repeat screening rounds ( year 3, 6, 9, 12 and 15).
  Distribution of PI-RADS (Prostate Imaging-Reporting and Data System; 1-5; 5=clinically significant cancer is highly likely to be present) scores among men undergoing an MRI

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Nordström, MD PhD, Principal Investigator — Karolinska Institutet
Locations (3):
- Sweden (3):
  - C-medical Odenplan Urology, Stockholm
  - Capio St Görans Hospital, Stockholm
  - Urologifocus, Stockholm

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nordstrom T, Picker W, Aly M, Jaderling F, Adolfsson J, Strom P, Haug ES, Eklund M, Carlsson S, Gronberg H. Detection of Prostate Cancer Using a Multistep Approach with Prostate-specific Antigen, the Stockholm 3 Test, and Targeted Biopsies: The STHLM3 MRI Project. Eur Urol Focus. 2017 Dec;3(6):526-528. doi: 10.1016/j.euf.2017.01.014. Epub 2017 Mar 28. PMID 28753850
- [Result] Nordstrom T, Discacciati A, Bergman M, Clements M, Aly M, Annerstedt M, Glaessgen A, Carlsson S, Jaderling F, Eklund M, Gronberg H; STHLM3 study group. Prostate cancer screening using a combination of risk-prediction, MRI, and targeted prostate biopsies (STHLM3-MRI): a prospective, population-based, randomised, open-label, non-inferiority trial. Lancet Oncol. 2021 Sep;22(9):1240-1249. doi: 10.1016/S1470-2045(21)00348-X. Epub 2021 Aug 13. PMID 34391509
- [Result] Eklund M, Jaderling F, Discacciati A, Bergman M, Annerstedt M, Aly M, Glaessgen A, Carlsson S, Gronberg H, Nordstrom T; STHLM3 consortium. MRI-Targeted or Standard Biopsy in Prostate Cancer Screening. N Engl J Med. 2021 Sep 2;385(10):908-920. doi: 10.1056/NEJMoa2100852. Epub 2021 Jul 9. PMID 34237810
- [Derived] Bjornebo L, Discacciati A, Falagario U, Vigneswaran HT, Jaderling F, Gronberg H, Eklund M, Nordstrom T, Lantz A. Biomarker vs MRI-Enhanced Strategies for Prostate Cancer Screening: The STHLM3-MRI Randomized Clinical Trial. JAMA Netw Open. 2024 Apr 1;7(4):e247131. doi: 10.1001/jamanetworkopen.2024.7131. PMID 38648061
- [Derived] Nordstrom T, Annerstedt M, Glaessgen A, Carlsson S, Clements M, Abbadi A, Gronberg H, Jaderling F, Eklund M, Discacciati A. Repeated Prostate Cancer Screening Using Prostate-Specific Antigen Testing and Magnetic Resonance Imaging: A Secondary Analysis of the STHLM3-MRI Randomized Clinical Trial. JAMA Netw Open. 2024 Feb 5;7(2):e2354577. doi: 10.1001/jamanetworkopen.2023.54577. PMID 38324313
- [Derived] Hao S, Heintz E, Ostensson E, Discacciati A, Jaderling F, Gronberg H, Eklund M, Nordstrom T, Clements MS. Cost-Effectiveness of the Stockholm3 Test and Magnetic Resonance Imaging in Prostate Cancer Screening: A Microsimulation Study. Eur Urol. 2022 Jul;82(1):12-19. doi: 10.1016/j.eururo.2021.12.021. Epub 2022 Jan 31. PMID 35094896
- [Derived] Nordstrom T, Jaderling F, Carlsson S, Aly M, Gronberg H, Eklund M. Does a novel diagnostic pathway including blood-based risk prediction and MRI-targeted biopsies outperform prostate cancer screening using prostate-specific antigen and systematic prostate biopsies? - protocol of the randomised study STHLM3MRI. BMJ Open. 2019 Jun 14;9(6):e027816. doi: 10.1136/bmjopen-2018-027816. PMID 31201191
- See also: Study homepage — http://sthlm3.se